CLINICAL TRIAL: NCT03658733
Title: Efficacy and Safety of a 14-day Modified Sequential Therapy for Refractory Helicobacter Pylori Infection: an Open Randomized Pilot Study
Brief Title: A Pilot Study of a 14-day Modified Sequential Therapy for Helicobacter Pylori Infection
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, director of Qilu Hospital gastroenterology department, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018SDU-QILU-G002
Record Dates: First submitted 2018-09-02; First posted 2018-09-05 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Helicobacter Pylori Infection
Keywords: Sequential therapy; Rescue treatment
MeSH Terms: interventions — Esomeprazole; Amoxicillin; Tetracycline; Furazolidone; Single Person; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Esomeprazole-containing therapy (Experimental): All the participants will go through a gastroscopy. Biopsy specimens will be taken for histologic assessment and rapid urease test. Two additional biopsy samples will be obtained from the antrum and body for bacterial culture and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment. Then, patients will receive a 14-day modified sequential therapy containing esomeprazole for the Helicobacter pylori eradication irrespective of antimicrobial susceptibility test results. The regimen contains esomeprazole, amoxicillin, tetracycline and furazolidone for the first 7 days, followed by esomeprazole,amoxicillin, tetracycline and colloidal bismuth pectin for the second 7 days.
  Drugs: 1. esomeprazole 40mg bid for 14 days, 2. amoxicillin 1000mg bid for 14 days, 3. tetracycline 500mg qid for 14 days, 4. furazolidone 100mg tid for the first 7 days, 5. colloidal bismuth pectin 200mg bid for the second 7 days.
  Interventions: Drug: esomeprazole, amoxicillin, tetracycline, furazolidone (only for the first 7 days), colloidal bismuth pectin (for the second 7 days)
- Rabeprazole-containing therapy (Active Comparator): All the participants will go through a gastroscopy. Biopsy specimens will be taken for histologic assessment and rapid urease test. Two additional biopsy samples will be obtained from the antrum and body for bacterial culture and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment. Then, patients will receive a 14-day modified sequential therapy containing rabeprazole for the Helicobacter pylori eradication irrespective of antimicrobial susceptibility test results. The regimen contains rabeprazole, amoxicillin, tetracycline and furazolidone for the first 7 days, followed by rabeprazole, amoxicillin, tetracycline and colloidal bismuth pectin for the second 7 days.
  Drugs: 1. rabeprazole 20mg bid for 14 days, 2. amoxicillin 1000mg bid for 14 days, 3. tetracycline 500mg qid for 14 days, 4. furazolidone 100mg tid for the first 7 days, 5. colloidal bismuth pectin 200mg bid for the second 7 days.
  Interventions: Drug: rabeprazole, amoxicillin, tetracycline, furazolidone (only for the first 7 days), colloidal bismuth pectin (for the second 7 days)

INTERVENTIONS:
Drug: esomeprazole, amoxicillin, tetracycline, furazolidone (only for the first 7 days), colloidal bismuth pectin (for the second 7 days) — Patients will go through a gastroscopy and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment. Then, patients will receive a 14-day modified sequential therapy containing esomeprazole for the Helicobacter pylori eradication. The regimen contains a double dose esomeprazole, amoxicillin, tetracycline and furazolidone for the first 7 days, followed by esomeprazole, amoxicillin , tetracycline and colloidal bismuth pectin for the second 7 days.
  Arms: Esomeprazole-containing therapy
Drug: rabeprazole, amoxicillin, tetracycline, furazolidone (only for the first 7 days), colloidal bismuth pectin (for the second 7 days) — Patients will go through a gastroscopy and antimicrobial susceptibility test. Liver and kidney function will be monitored by blood test before and after the treatment. Then, patients will receive a 14-day modified sequential therapy containing rabeprazole for the Helicobacter pylori eradication. The regimen contains a double-dose rabeprazole, amoxicillin, tetracycline and furazolidone for the first 7 days, followed by rabeprazole, amoxicillin , tetracycline and colloidal bismuth pectin for the second 7 days.
  Arms: Rabeprazole-containing therapy

SUMMARY:
The purpose of this study is to assess efficacy of a new 14-day sequential therapy for the rescue treatment of refractory Helicobacter pylori infection, and whether it is safe while maintaining an ideal eradication rates. The researchers also want to testify whether a double-dose rabeprazole has equal efficacy to double-dose esomeprazole to provide sufficient acid inhibition.

DETAILED DESCRIPTION:
Half of the world's population is infected with Helicobacter pylori. Strong evidence supports that H.pylori eradication is an effective approach to reduce the risk of developing gastric cancer. However, eradication rates of first-line therapy decreased over years due to the rapidly emerging antibiotic resistance of H. pylori worldwide. An ideal rescue therapeutic regimen to cure refractory H.pylori infection is currently warranted. Traditional sequential therapy failed to achieve an ideal eradication rates (over>95%) as a third line treatment in the region with high antibiotic resistance. This study aims to evaluate the efficacy of 14-day modified sequential therapy in the patients with two or more treatment failure, and whether the adverse effects of this new modified sequential therapy are tolerable. Then, this study will also compare the performance of a double-dose esomeprazole with double-dose rabeprazole containing therapy to optimize therapeutic regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-70 with persistent H. pylori infection.
* Patients failed at least three different standard eradication therapies before. Previous standard eradication therapy was defined as a 10-day or 14-day quadruple regimen designed according to Maastricht V report.

Exclusion Criteria:

* Patients unable or unwilling to receive gastroscopy.
* Patients treated with H2-receptor antagonist, PPI, bismuth and antibiotics in the previous 4 weeks.
* Patients with gastorectomy, acute GI bleeding and advanced gastric cancer.
* History of allergy to any of the drugs used in the study.
* Severe concomitant cardiovascular, respiratory, or endocrine diseases, clinically significant renal or hepatic disease, hematologic disorders and any other clinically significant medical condition that could increase risk.
* Currently pregnant or lactating.
* Severe neurologic or psychiatric disorders.
* Alcohol abuse or drug addiction.
* Patients with compliance lower than 90% in any previous treatment are not included.
* Inability to provide informed consent and other situations that could interfere with the examination or therapeutic protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rates | 6 months
  Both intention to treat(ITT) and per-protocol(PP) analyses will be used for the assessment of the eradication rates of Helicobacter pylori infection. The ITT analysis includes all randomly assigned patients who take at least one dose of the study medications. The PP analysis is limited to patients who take over 90% of the study medications and complete follow-up.

SECONDARY OUTCOMES:
The rate of adverse events happening | 6 months
  Parameters of liver and kidney function before and after the treatment will be compared. Common adverse events will be measured and patients will rate the severity of their symptoms from 0 (none) to 8 (severe) points during the treatment process.
The change of dyspepsia symptoms after Helicobacter pylori eradication | 6 months
  Dyspepsia symptoms will be recorded before and after the treatment. Patients will rate the severity of their symptoms from 0 (none) to 8 (severe) points.
The rate of good compliance | 6 months
  Patients taken over 90% of drugs are considered to have a good compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Xiuli Zuo, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu J, Ji CR, Li YY, Qiao C, Hu JN, Wan M, Lin MJ, Lin BS, Wang J, Zha J, Li LX, Zuo XL. Two Different 1-Week Quadruple Therapies Given Back-to-Back Consecutive Therapy for Difficult-to-Treat Helicobacter pylori Infection: A Pilot Study. Clin Transl Gastroenterol. 2021 Aug 16;12(8):e00391. doi: 10.14309/ctg.0000000000000391. PMID 34397042